CLINICAL TRIAL: NCT03188991
Title: A Trial Evaluating Escalating Doses and the Safety of Intracystic Injection of NanoPac® in Subjects With Mucinous Cystic Pancreatic Neoplasms
Brief Title: Intracystic Injection of NanoPac® in Subjects With Mucinous Cystic Pancreatic Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2017-01
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Mucinous-Cystic Neoplasm
Keywords: pancreatic cystic neoplasm; pancreatic cyst; pancreatic mucinous cyst; pancreatic neoplasms; digestive system neoplasms; pancreatic diseases; mucinous cystic neoplasm
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms; Digestive System Neoplasms; Pancreatic Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, dose rising trial. During the dose escalation phase, subjects will be enrolled in sequential cohorts of NanoPac®. Each cohort will have three subjects, with cohorts enrolled sequentially starting at the lowest concentration. Following DSMB review of the cohort data, the next cohort may begin enrolling, an additional three subjects at the current dose may be enrolled, or, if the first dose does not provide adequate safety and tolerability, the study may be halted. The dose determined to be the most suitable for further evaluation, defined as the highest dose with an acceptable safety and tolerability profile (as determined by the DSMB), will be the dose used in the second phase of the study which will enroll 9 additional subjects. Subjects enrolled in the second phase of the study will also receive a second injection of NanoPac at the same dose 12 weeks after the first NanoPac injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: NanoPac® 6 mg/mL (Experimental): Single intracystic injection of NanoPac® at a dose of 6 mg/mL in a volume sufficient to fill the cyst, at least equal to the amount of cyst fluid aspirated
  Interventions: Drug: NanoPac®
- Dose Escalation: NanoPac® 10 mg/mL (Experimental): Single intracystic injection of NanoPac® at a dose of 10 mg/mL in a volume sufficient to fill the cyst, at least equal to the amount of cyst fluid aspirated
  Interventions: Drug: NanoPac®
- Dose Escalation: NanoPac® 15 mg/mL (Experimental): Single intracystic injection of NanoPac® at a dose of 15 mg/mL in a volume sufficient to fill the cyst, at least equal to the amount of cyst fluid aspirated
  Interventions: Drug: NanoPac®
- Second Phase: NanoPac® at Best Dose (Experimental): Intracystic injection of NanoPac®. The dose administered in the second phase will be determined during the dose escalation phase. Subjects will receive two NanoPac® injections, with the second injection administered 12 weeks after the first injection.
  Interventions: Drug: NanoPac®

INTERVENTIONS:
Drug: NanoPac® — NanoPac® (Sterile Nanoparticulate Paclitaxel) for intracystic injection via endoscopic ultrasound-guided injection (EUS-FNI)

SUMMARY:
This study will evaluate intracystic NanoPac® (Sterile Nanoparticulate Paclitaxel) administered via endoscopic ultrasound-guided fine needle injection (EUS-FNI) in subjects with mucinous cystic pancreatic neoplasms.

DETAILED DESCRIPTION:
In this open-label, dose rising trial, subjects with mucinous cystic pancreatic neoplasms will receive intracystic NanoPac® via endoscopic ultrasound-guided fine needle injection (EUS-FNI).

In the dose escalation phase, subjects will be enrolled in sequential cohorts of NanoPac® at 6, 10, and 15 mg/mL at volumes sufficient to fill the cyst, at least equal to the amount of cyst fluid aspirated. Each cohort will have three subjects, with cohorts enrolled sequentially starting at the lowest concentration. Following Data Safety Monitoring Board (DSMB) review of the cohort data, the next cohort may begin enrolling, an additional three at the current dose may be enrolled, or if the first dose does not provide adequate safety and tolerability the study may be halted. The dose determined to be the most suitable for further evaluation, defined as the highest dose with an acceptable safety and tolerability profile (as determined by the DSMB), will be the dose used in the second phase of the study which will enroll 9 additional subjects. Subjects enrolled in the second phase of the study will also receive a second injection of NanoPac at the same dose 12 weeks after the first NanoPac injection..

Plasma samples will be taken on the day(s) of NanoPac® injection at 1 and 2 hours after injection, as well as at each of the subsequent study visits, to characterize the pharmacokinetics (PK) of intracystic NanoPac®.

Subjects will be followed for 6 months after the first NanoPac® injection for safety, tolerability and cyst response to therapy (as shown by imaging).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Patients over the age of 18;
* Recently confirmed mucinous cystic pancreatic neoplasm; may be confirmed by presence of mucin, cyst fluid carcinoembryonic antigen (CEA) above 192 U/L, or other reliable diagnostic means such as endomicroscopy; KRAS analysis may also be performed at the discretion of the Investigator;
* Unilocular cyst with diameter of at least 1.5 cm but no more than 4 cm;
* Normal hematologic, hepatic, and renal function at study entry;
* Appropriate steps taken to minimize or avoid the potential for pregnancy for subjects of child-bearing potential.*

  * Note: A female patient is considered to be of childbearing potential unless she has had a hysterectomy, is at least one year postmenopausal or has undergone tubal ligation. For the purposes of this study, adequate birth control includes at least one medically approved and highly effective method of birth control, defined as those which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly, such as implants, injectables and oral contraceptives combined with the use of condoms. Only male patients whose vasectomy has been confirmed by semen analysis at least 3 months after the vasectomy are allowed not to use acceptable contraceptive methods.

Exclusion Criteria:

* Positive cytology indicating malignancy;
* Thrombotic or embolic events;
* Known hypersensitivity to study agent;
* Known drug or alcohol abuse;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Second Phase: NanoPac® 15 mg/mL (Up to Two Injections): Intracystic injection of NanoPac®. The dose administered in the second phase will be determined during the dose escalation phase. Subjects will receive up to two NanoPac® injections, with the second injection administered 12 weeks after the first injection.
  NanoPac®: NanoPac® (Sterile Nanoparticulate Paclitaxel) for intracystic injection via endoscopic ultrasound-guided injection (EUS-FNI)
Period: Overall Study
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections)
Started | 3 | 3 | 3 | 11
Completed | 3 | 3 | 3 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects (n=20) who received at least one NanoPac injection (n=19) were designated as the Safety Population, and included in the analysis population for all outcome analyses. The subject who withdrew consent prior to any NanoPac treatment is not included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.3) | 73.7 (11.5) | 59.7 (9.1) | 67.8 (6.6) | 67.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 6 | 13
  Male | 0 | 1 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 3 | 3 | 3 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 1 | 3 | 3 | 8 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Body Mass Index (BMI) (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 34.83 (11.71) | 27.93 (10.20) | 26.67 (3.43) | 32.82 (7.17) | 31.39 (7.91)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Treatment Emergent Adverse Events will include laboratory assessments, physical examination findings, and vital signs.
Time Frame: Up to 6 (six) months after first NanoPac® injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections)
Number analyzed (Participants) | 3 | 3 | 3 | 10
Participants | 3 | 3 | 3 | 9

2. Secondary Outcome: Cyst Volume Response
Description: Cyst volume at screening will be compared with the volume at Weeks 12 and 24 (or early termination).
Time Frame: Screening and 6 (six) months after first NanoPac® injection
Population: In the dose escalation phase, baseline imaging data for the measurement of cyst diameters and calculation of cyst volume was available in all subjects. At Week 12, 18 of 19 subjects had three cyst diameters available for analyses. At Week 24, 17 of 19 subjects had three cyst diameters available for analyses.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections)
Number analyzed (Participants) | 3 | 3 | 3 | 10
mL
  Screening | 7.770 (3.283) | 4.810 (5.109) | 10.960 (8.484) | 11.442 (8.132)
  Week 12 | 5.710 (3.892) | 3.453 (2.188) | 9.633 (9.284) | 12.293 (10.755)
  Week 24/EOS | 4.140 (3.920) | 4.383 (0.521) | 8.533 (7.183) | 11.138 (11.931)

ADVERSE EVENTS:
Time Frame: AEs were collected at all study visits from the time of dosing (Day 1 through Week 24).
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 3/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: NanoPac® 6 mg/mL (N=3) | Dose Escalation: NanoPac® 10 mg/mL (N=3) | Dose Escalation: NanoPac® 15 mg/mL (N=3) | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections) (N=10)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: NanoPac® 6 mg/mL (N=3) | Dose Escalation: NanoPac® 10 mg/mL (N=3) | Dose Escalation: NanoPac® 15 mg/mL (N=3) | Second Phase: NanoPac® 15 mg/mL (Up to Two Injections) (N=10)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Duodenal ulcer, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI Motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Hernia pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
URTI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infec. (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WBC count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03188991/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT03188991/SAP_001.pdf